CLINICAL TRIAL: NCT06952101
Title: INTERPRETE: a Global, Integrated, Personalized, Stage-related, Multimodal Therapeutic Approach for Rectal Adenocarcinoma Based on Organ Sparing and Mininvasivity
Brief Title: A Global, Integrated, Personalized, Stage-related, Multimodal Therapeutic Approach for Rectal Adenocarcinoma Based on Organ Sparing and Mininvasivity
Acronym: INTERPRETE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-FPO24
Record Dates: First submitted 2025-02-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Rectal Adenocarcinoma; Non Metastatic
Keywords: Rectal Adenocarcinoma; mininvasivity; organ sparing; surgical rectal resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sparing Approach (Experimental): Group 1 - Patients with high-risk pT1cN0M0 cancerized adenoma, diagnosed through histological analysis following Endoscopic Resection (ER) or Local Excision (LE).
  For patients classified as "high-risk" pT1 at final pathology, an experimental sparing strategy is proposed, consisting of experimental chemoradiotherapy (spCRT) followed by a Watch and Wait (W&W) approach (also referred to as Organ-Sparing Approach, OSA), in selected cases.
  Interventions: Procedure: Sparing Approach
- Experimental Chemoradiotherapy: A Path to Conservative Treatment (Experimental): Group 2 - Patients with cT2N0 tumors, typically candidates for upfront radical rectal resection. An alternative, non-operative approach is proposed based on experimental chemoradiotherapy (spCRT).
  According to current literature, the pathologic Complete Response (pCR) rate following CRT significantly exceeds the 25% commonly reported for intermediate to advanced rectal tumors. Clinical Complete Response (cCR) or clinical Minimal Residual disease (cMR) will be assessed through multidisciplinary, high-resolution restaging, including:
  Pelvic Magnetic Resonance Imaging (MRI) Positron Emission Tomography (PET) Thoraco-abdominal Computed Tomography (CT) Endorectal Ultrasound (ERUS) Rectoscopy
  In patients achieving cCR or cMR, a Watch & Wait (W&W) strategy or Local Excision/Transanal Minimally Invasive Surgery (LE/TAMIS) may be proposed to avoid the physical and psychological burden of major surgery. An intensive follow-up protocol will be implemented.
  Interventions: Procedure: experimental chemoradiotherapy
- tandard Chemotherapy Approach: Restaging for Conservative Surgery (Active Comparator): Group 3 - Patients with cT3-4, N+, CRM-positive, or EMVI-positive tumors will receive standard chemoradiotherapy (stCRT) as the initial treatment.
  Patients achieving cCR or cMR at restaging will be evaluated for organ-sparing strategies, including Watch & Wait (W&W) or LE/TAMIS, in accordance with existing multicenter clinical research protocols. In cases where a conservative approach is not feasible, standard surgical treatment will follow.
  Interventions: Procedure: Standard Chemotherapy

INTERVENTIONS:
Procedure: Sparing Approach — Accurate staging with Pelvic MRI, CT scan, PET total body have to be performed before local excision in order to exclude false positive mesorectal lymph nodes. Subsequent Wait and See (W&S) approach could be proposed.
  Arms: Sparing Approach
Procedure: experimental chemoradiotherapy — Participants with cT2N0 rectal tumors are typically candidates for upfront surgical resection. The investigators propose an alternative approach based on experimental chemoradiotherapy (spCRT). Literature suggests that pathologic complete response (pCR) rates after CRT are significantly higher than the 25% described for intermediate-advanced tumors. The investigators will assess clinical complete response (cCR) or complete metabolic response (cMR) through a multidisciplinary restaging process, including MRI, PET, thorax-abdomen CT scan, ERUS, and rectoscopy. In participants achieving cCR or cMR, a Watch and Wait (W&S) strategy or Local Excision/Transanal Minimally Invasive Surgery (LE/TAMIS) may be proposed to avoid the physical and psychological consequences of major surgery, followed by a rigorous surveillance program.
  Arms: Experimental Chemoradiotherapy: A Path to Conservative Treatment
Procedure: Standard Chemotherapy — Tumors will be initially treated with standard CRT (stCRT). Patients who reach cCR-cMR at restaging they are already candidates to sparing approaches with W&S/LE/TAMIS according to Multicentric Resarch Study Protocol
  Arms: tandard Chemotherapy Approach: Restaging for Conservative Surgery

SUMMARY:
A phase II, single-center, non-profit, interventional study on patients affected by rectal adenocarcinoma. Patients will be stratified into three groups based on pre-treatment clinical stage. The study investigates and may propose a comprehensive, stage-specific, multimodal approach to rectal adenocarcinoma, with a focus on organ preservation even in early stages (cT1-2N0). When organ-sparing strategies are not feasible, the approach prioritizes minimally invasive techniques (laparoscopic and robotic) to reduce the physical, psychological, and quality-of-life impact on patients.

DETAILED DESCRIPTION:
Patients affected by rectal adenocarcinoma will be stratified into three groups according to pre-treatment clinical stage:

Group 1: pT1cN0M0 tumors may be candidates for Endoscopic Resection (ER), Local Excision (LE), or TransAnal Minimally Invasive Surgery (TAMIS). If final pathology classifies these tumors as "high-risk" pT1, patients are typically candidates for radical rectal resection due to an estimated 20% risk of mesorectal lymph node metastases. However, many patients refuse surgery and opt for direct follow-up despite the increased risk of recurrence. The investigators propose an alternative treatment with experimental chemoradiotherapy (spCRT) to reduce the risk of local relapse in patients unwilling to undergo surgery, followed by an intensive surveillance protocol. Accurate staging with pelvic MRI, CT scan, and whole-body PET must be performed prior to local excision to exclude false-positive mesorectal lymph nodes. A subsequent Watch and Wait (W&S) strategy may be considered.

Group 2: cT2N0 tumors are typically managed with upfront surgical rectal resection. This study proposes an alternative approach based on spCRT. Literature indicates that the rate of pathological Complete Response (pCR) after CRT is significantly higher than the 25% typically reported for intermediate to advanced rectal tumors. Clinical Complete Response (cCR) or clinical Minimal Residual disease (cMR) will be assessed through multidisciplinary, high-resolution restaging including pelvic MRI, whole-body PET, thoraco-abdominal CT scan, EndoRectal Ultrasound (ERUS), and rectoscopy. In patients achieving cCR or cMR, a W&S approach or LE/TAMIS may be proposed to minimize the psychological and physical burden of surgery, with subsequent close surveillance.

Group 3: Patients with cT3-4, N+, circumferential resection margin positive (CRM+), or extramural vascular invasion (EMVI+) tumors will initially receive standard chemoradiotherapy (stCRT). Those who achieve cCR or cMR at restaging may be considered for organ-sparing approaches (W&S/LE/TAMIS) according to established multicenter research protocols.

All patients in Group 1 and Group 2 who do not achieve cCR or cMR will be managed according to the principle of minimal invasiveness. These patients will undergo laparoscopic or robotic rectal resection with preservation of pelvic autonomic nerves, aimed at reducing genitourinary dysfunction and improving short-term outcomes (e.g., reduced postoperative pain, fewer abdominal wall hernias, faster bowel function recovery, and quicker return to daily activities). Recovery will be further optimized through integration with Enhanced Recovery After Surgery (ERAS) protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 yrs old
* Patients able to sign the informed consent
* Patients with High Risk pT1 rectal adenocarcinoma endoscopically excised
* Patients with cT2-3aN0 rectal adenocarcinoma who has complete/major response to EXPERIMENTAL CRT
* Patients with cT3b4N0-1 rectal adenocarcinoma who has complete/major response to STANDARD CRT

Exclusion Criteria:

* cT2-4 any NM0 who don't reach cCR or cMR after experimental/standard CRT
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and Validation of a Clinical-Radiologic-Molecular Scoring System for Predicting Pathologic Complete Response (pCR) in Rectal Cancer | 4 Years
  Quantification of the probability of achieving pathologic complete response (pCR) following chemoradiotherapy (CRT) through a composite scoring system integrating:
  Radiomic data from Pelvic MRI and PET Endoscopic findings (e.g., mucosal healing, residual lesion) Molecular markers (e.g., Microsatellite Instability [MSI], mutations in BER, SSB, and NER DNA repair pathways).
  Scoring Output: Probability value (0-1) or risk class (low, intermediate, high) for likelihood of pCR.
  Purpose: Stratify patients into low- or high-probability groups to support treatment decision-making (e.g., immediate surgery vs. organ-sparing strategies).

SECONDARY OUTCOMES:
Success Rate of the Organ Sparing Approach (OSA) | 4 Years
  Percentage of patients undergoing OSA who achieve a positive clinical response (defined as clinical complete response or stable disease without need for radical resection).
  Assessment Method: Clinical examination, imaging (MRI, PET), histological evaluation, and follow-up data.
  Unit of Measure: Percentage (%) of responders
Long-Term Disease-Free Survival in Patients Undergoing Organ Sparing Approach (OSA) vs. Radical Surgical Resection (RSR) | 5 Years
  Comparison of local and distant recurrence rates between OSA and RSR groups.
  Assessment Tools:
  Proctoscopy Pelvic MRI CT scan of thorax and abdomen Whole-body PET Unit of Measure: Percentage (%) of patients without recurrence
  Definition of Outcome: Disease-free survival at 3 and 5 years post-treatment.
Short-Term General Cancer-Related Quality of Life (QoL) in OSA vs. Resection Groups | Baseline (before CRT), Post-CRT, Post-surgery, 6-month follow-up, 12-month follow-up
  Evaluation of patient-reported general cancer-related quality of life using the EORTC QLQ-C30 questionnaire. Scores range from 0 to 100, with higher scores indicating better functioning.
  Measure: Units on EORTC QLQ-C30 scale (0-100)
Short-Term Colorectal Cancer-Specific Functioning in OSA vs. Resection Groups | Baseline (before CRT), Post-CRT, Post-surgery, 6-month follow-up, 12-month follow-up
  Evaluation of patient-reported colorectal cancer-specific functioning using the EORTC QLQ-CR38 questionnaire. Scores range from 0 to 100, with higher scores indicating better quality of life.
  Measure:
  Units on EORTC QLQ-CR38 scale (0-100)
Bowel Dysfunction After Rectal Surgery (Low Anterior Resection Syndrome - LARS) in OSA vs. Resection Groups | Baseline (before CRT), Post-CRT, Post-surgery, 6-month follow-up, 12-month follow-up
  Assessment of bowel dysfunction after rectal surgery using the Low Anterior Resection Syndrome (LARS) Score. Scores range from 0 to 42, with higher scores indicating worse function.
  Measure:
  Units on LARS Score scale (0-42)

CONTACTS AND LOCATIONS:
Overall Officials: Felice Borghi, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Department of Surgical Oncology - FPO-IRCCS Institute for Cancer Research and Treatment, Candiolo, Turin, Italy

IPD SHARING:
Plan to Share IPD: No